CLINICAL TRIAL: NCT02088320
Title: Measurement of Pulmonary Transit Time by Echocardiography: Comparison With Cardiac MRI
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Kenneth Monahan, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 131355
Record Dates: First submitted 2014-03-10; First posted 2014-03-14 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Patients Undergoing Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The focus of the present study is to further develop an echocardiographic technique to measure cardiopulmonary transit time (PTT) and pulmonary blood volume (PBV) using ultrasound contrast.

The Specific Aims for the present study are as follows:

1. To compare echocardiography-based PTTs and cardiac MRI-based PTTs obtained using a 'peak-to-peak' method
2. To further quantify the relationship between echocardiographically-derived PTT, using Optison, and existing echocardiographic methods used to determine ventricular function
3. To measure the reproducibility of echocardiographically-based PTT using Optison.

DETAILED DESCRIPTION:
Study Procedures The measurement of PTT and PBV has been described in detail in our prior protocol. These calculations and techniques are identical for the current study. In addition, we may place additional regions of interest (ROIs) during the off-line analysis, but this step would not influence the data acquisition during the TEE or the TEE procedure itself.

Note that placement of a peripheral intravenous (IV) catheter is standard-of-care for patients undergoing a TEE.

Acquisition and Analysis of Data:

The following is the anticipated flow of data acquisition and analysis:

1. Prior to or upon arrival to the TEE Suite, prospective patients will be screened by study personnel for informed consent.
2. After informed consent is obtained, the patient will undergo a focused TTE in the TEE Holding Room prior to the TEE. One or two doses of echocardiographic contrast will be administered to obtain PTT via TTE to facilitate comparison to PTT derived from TEE (Specific Aim #3). Prior to ultrasound contrast administration, an agitated saline injection will be given if intra-cardiac shunt is suggested by color Doppler evaluation. If a shunt is present, contrast would not be administered and the patient would be unenrolled from the study.
3. During the TEE, under direct supervision of an attending cardiac anesthesiologist and/or an attending cardiologist, up to 2 additional doses of echocardiographic contrast would be administered. A sub-set of patients will receive 2 doses to facilitate comparison of PTT obtained from different views (Specific Aim #2). This is analogous to our previous protocol in which multiple doses of contrast are administered in order to assess reproducibility of PTT measurements.
4. As part of standard-of-care, all patients that have completed a TEE are monitored in the TEE Suite for at least 30 minutes including assessment of blood pressure, heart rate, and oximetry.

Studies to be analyzed will be locked on the Echocardiography cart and the data will be transmitted to a separate work-station for 'off-line' analysis using dedicated software. As a back-up, the data will also be stored on DVDs, which will be stored under lock and key in the PI or co-investigator's offices in VHVI. As described in our prior protocol, clinical and echocardiographic data will be entered into a REDCap database.

We estimate that conducting the limited TTE prior to the scheduled TEE will take ~ 10-15 minutes. However, these steps can be carried out in the TEE Holding Room while another patient is getting a TEE in the Procedure Room and should therefore not add procedural or waiting time to the length of the scheduled TEE. If the first TEE patient of the day is enrolled in the study, study personnel can perform the TTE portion as the Procedure Room is being prepped for the TEE.

During the TEE, administration of contrast in the manner described above is estimated to add ~ 10-15 minutes to the duration of the procedure. This includes administration of the contrast and, in the case of administering multiple doses, waiting for the initial contrast injection to wash out, and then administering an additional dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female sex, age >18 years who are having an echocardiogram done for clinical reasons. Based on the potential for further support of our work, this may expand to include volunteers who would otherwise not be undergoing an echocardiogram.
2. Negative pregnancy test for women of childbearing potential
3. If eligible for cMRI, estimated glomerular filtration rate (eGFR) of > 30 mL/min
4. If eligible for cMRI, cMRI checklist obtained
5. Able to give informed consent

Exclusion Criteria:

1. Unable to give informed consent
2. Known right-to-left, bidirectional, or transient right-to-left cardiac shunts
3. Currently participating in another clinical treatment trial
4. Known allergic reaction to Optison ultrasound contrast
5. If eligible for cMRI, known allergic reaction to cMRI contrast
6. If eligible for cMRI, contraindication to cMRI
7. If eligible for cMRI, pre-cMRI eGFR < 30 mL/min
8. Pregnancy/Nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female sex, age >18 years who are having an echocardiogram done for clinical reasons.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-06-26 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
1. To compare echocardiography-based PTTs and cardiac MRI-based PTTs obtained using a 'peak-to-peak' method | This will be assessed at the study visit. This study only have one study visit per patient.

SECONDARY OUTCOMES:
2. To further quantify the relationship between echocardiographically-derived PTT, using Optison, and existing echocardiographic methods used to determine ventricular function | This will be assessed at the study visit. This study only have one study visit per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Monahan, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States